CLINICAL TRIAL: NCT06878950
Title: The GAIN Study: The Gastroschisis And Early Infant Nutrition Study
Brief Title: Early Feeds in Gastroschisis
Acronym: GAIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: The Gerber Foundation (Other); University of California, Los Angeles (Other); University of California Fetal Consortium (Unknown); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2216195; UL1TR001860 (NIH)
Record Dates: First submitted 2025-03-04; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Gastroschisis
Keywords: Gastroschisis; Early feeds in Gastroschisis
MeSH Terms: conditions — Gastroschisis

STUDY DESIGN:
Intervention Model Description: The study evaluates the feasibility and safety of a standardized early feeding protocol for neonates with presumed simple gastroschisis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Early Feeding Protocol Group (Experimental): This arm involves neonates with presumed simple gastroschisis who will be subjected to an early feeding protocol. The protocol specifies initiating human milk feeds within 48 hours of surgical repair of gastroschisis. Feeds are advanced based on tolerance and clinical assessment, with a focus on promoting oral motor skill development.
  Interventions: Procedure: Early Feeding Protocol

INTERVENTIONS:
Procedure: Early Feeding Protocol — The intervention includes removal of Replogle within 24 hours of abdominal closure and the initiation of introductory feeds within 48 hours of abdominal closure.
  Other Names: Early Initiation of Human Milk Feeds

SUMMARY:
This study aims to evaluate the feasibility of initiating early feeds in neonates with gastroschisis, a condition where infants are born with their intestines outside the body.

ELIGIBILITY:
Inclusion Criteria:

* Neonates with presumed simple gastroschisis
* Born at ≥ 34 weeks' gestation
* Hemodynamically stable
* Consented within 48 hours after abdominal closure
* Mothers who are ≥16 years old
* Mothers who speak English or Spanish

Exclusion Criteria:

* Neonates with evidence of complex gastroschisis at time of closure (any ischemic bowel, intestinal perforation, or obvious atresia with mesenteric defect)
* Presence of any major congenital anomalies
* Neonates who are receiving ionotropic medications
* Neonates who are wards of the state
* Neonates whose care is considered to be futile or those undergoing re-direction of care
* Neonates participating in another interventional trial
* Any patient deemed unfit for participation by study investigator(s)

Ages: 0 Days to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Enrollment in Early Feeding Study Cohort | From prenatal period within the first 24 hours of abdominal closure
  Proportion of eligible neonates with gastroschisis whose parents/guardians consent to enrollment in the study.

SECONDARY OUTCOMES:
Feasibility of Protocol Adherence | From abdominal closure to 48 hours after closure.
  Proportion of enrolled neonates who are initiated on introductory feeds within 48 hours of abdominal closure.
Fidelity to Protocol | From abdominal closure through discharge from the hospital, average of 90 days
  Proportion of enrolled infants with gastroschisis who adhere to the remainder of the protocol without major deviations. Feasibility will be assessed using protocol adherence tracking forms completed by study team.
Protocol Withdrawal Rate | From time of enrollment (prenatal) to hospital discharge, an average of 90 days
  Proportion of enrolled infants who withdraw from the study

OTHER OUTCOMES:
Outcomes of of Adverse Events | From enrollment through hospital discharge, an average of 90 days
  This exploratory outcome is measuring the incidence of severe adverse events in neonates enrolled in the early feeding protocol study.
  Adverse events include:
  * Necrotizing enterocolitis (>Stage II)
  * Sepsis
  * Abdominal compartment syndrome
  * Additional abdominal surgeries (excluding primary closure)
  * Mortality
Outcomes of Hospital Admission Duration | From birth admission to hospital through discharge, assessed up to 1 year
  This exploratory outcome measures the total duration of length (days) of hospital stay.
Outcome of Duration of Parenteral Nutrition | From initiation of parenteral nutrition through achievement of enteral autonomy, assessed up to 1 year
  This exploratory outcome measures the total duration of parenteral nutrition (days) in enrolled patients.
Outcome of Feeding Progression | From initiation of feeds through achievement of enteral autonomy, assessed up to 1 year
  This exploratory outcome measures the feeding progression (time to first feed (days) and time to full feeds (days)) in infants enrolled.
Outcome of Growth Parameters | From birth admission to hospital through discharge, assessed up to 1 year
  This exploratory outcomes measures the changes in growth parameters (height, weight) using calculated z-scores (as measured by standard deviations from the mean, presented in percentages relative to average for age).
Feasibility of Data Collection of Direct Breastfeeding Practices | Assessed from birth through hospital discharge, an average of 90 days
  Assessment of the feasibility of obtaining information related to breastfeeding practices through electronic medical records, using dichotomous measures of whether parent had direct breastfeeding during hospitalization and at time of discharge (48 hours prior to hospital discharge).

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Cacho, DO, Principal Investigator — University of California, Davis; Geoanna Bautista, MD, Principal Investigator — University of California, Davis
Locations (2):
- United States (2):
  - University of California Los Angeles, Los Angeles, California
  - UC Davis Children's Hospital, Sacramento, California

IPD SHARING:
Plan to Share IPD: Yes
After the primary study results are published, individual participant data will be de-identified and made available to qualified researchers upon request, subject to a data use agreement and review by the study team. Access will be granted within 12 months of a successful application, provided the request aligns with the study's scientific objectives, the intended study is IRB approved and adheres to ethical data protection guidelines.
Supporting Information: Study Protocol, ICF
Time Frame: Starting 6 months after publication
Access Criteria: The study team will review application requests submitted by interested researchers. The intended study must align with our study's scientific objectives, be IRB approved, and adhere to ethical data protection guidelines.

REFERENCES:
- [Background] Hobson D, Spence K, Trivedi A, Thomas G. Differences in attitudes to feeding post repair of Gastroschisis and development of a standardized feeding protocol. BMC Pediatr. 2019 Dec 4;19(1):475. doi: 10.1186/s12887-019-1858-z. PMID 31801489
- [Background] DeUgarte DA, Calkins KL, Guner Y, Kim J, Kling K, Kramer K, Lee H, Lusk L, Saadai P, Uy C, Rottkamp C; University of California Fetal Consortium. Adherence to and outcomes of a University-Consortium gastroschisis pathway. J Pediatr Surg. 2020 Jan;55(1):45-48. doi: 10.1016/j.jpedsurg.2019.09.048. Epub 2019 Oct 27. PMID 31704046
- [Background] Jyoti J, James-Nunez K, Spence K, Parkinson B, Thomas G, Trivedi A. Evaluation of gastroschisis feeding protocol: A retrospective cohort study. J Paediatr Child Health. 2024 Nov;60(11):675-679. doi: 10.1111/jpc.16657. Epub 2024 Aug 29. PMID 39206671